CLINICAL TRIAL: NCT01637701
Title: Comparison of Pasmakinetic Enucleation of the Prostate With Bipolar Transurethral Resection of the Prostate for the Treatment of Benign Prostatic Hypertrophy Patients With Large Prostate
Brief Title: Plasmakinetic Enucleation of the Prostate to Treat Benign Prostatic Hypertrophy Patients With Large Prostate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fuzhou General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PkEP-TURP-2004
Record Dates: First submitted 2012-07-04; First posted 2012-07-11 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-07

CONDITIONS: BPH With Large Prostate
Keywords: benign prostatic hypertrophy; bipolar transurethral resection of the prostate; plasmakinetic enucleation of the prostate
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PkEP (Active Comparator): Patients in this group undergo PkEP using the Gyrus plasmakinetic tissue management system (Gyrus Medical Ltd,Bucks,UK).
  Interventions: Procedure: PkEP
- B-TURP (Active Comparator): Patients in this group undergo B-TURP using the Gyrus plasmakinetic tissue management system (Gyrus Medical Ltd,Bucks,UK).
  Interventions: Procedure: B-TURP

INTERVENTIONS:
Procedure: PkEP — Plasmakinetic enucleation of the prostate
  Arms: PkEP
Procedure: B-TURP — Bipolar transurethral resection of the prostate
  Arms: B-TURP

SUMMARY:
The goal of this study is to compare the perioperative and postoperative characters of plasmakinetic enucleation of the prostate(PkEP) with bipolar TURP(B-TURP) for BPH patients with large prostate.

DETAILED DESCRIPTION:
Despite the availability of numerous minimally invasive alternatives, monopolar transurethral resection of the prostate (TURP) remains the most frequently performed operation for benign prostatic hypertrophy (BPH) with small to moderate size prostates. Nevertheless, TURP for large prostates is associated with various complications and unsatisfactory long-term results. B-TURP and PkEP have both been proved to have more favorable postoperative outcomes than monopolar TURP. But whether B-TURP or PkEP is better remain controversial. We aim to compare the perioperative and postoperative characters of PkEP with B-TURP for BPH patients with large prostate. Moreover, we evaluate the long-term results of both approaches.

ELIGIBILITY:
Inclusion Criteria:

* Qmax < 10 mL/s, IPSS >19
* Age between 50 and 70 years
* Prostate volume between 70 and 200 mL, as determined by TRUS, and medical therapy failure.

Exclusion Criteria:

* Patients with neurogenic bladder
* Urethral stricture
* Bladder tumor
* Prostate cancer and previous prostate bladder neck
* Urethral surgery
* PSA>4ng/ml, or receiving prostate biopsy within 3 months

Ages: 50 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2004-06; Primary Completion 2006-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
time of catheterization
  At the end of both procedures, a 22F three-way Folley catheter was inserted and continuous bladder irrigation was performed. Irrigation was discontinued when the catheter drainage became clear, and the catheter was removed 6 h later.Two experienced urologists who were unaware of the surgical modality used decided bladder irrigation and catheter removal for all cases.

SECONDARY OUTCOMES:
Operation time
resected adenoma weight as a measure of treatment efficacy
changes in serum haemoglobin as a measure of one of the complications
postoperative International Prostate Symptom Score as a measure of treatment efficacy and durability | 5 years
postoperative Qmax as a masure of treatment efficacy and durability | 5 years
re-operation rate as a measure of durability | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jianming Tan, M.D. & Ph.D., Study Director — Fuzhou General Hospital
Locations (1):
- Fuzhou General Hospital, Fuzhou, Fujian, China